# The ARMOR Trial Commensal Oral Microbiota as a Trigger of Oral Mucositis Severity

**NIDCR Protocol Number: 18-042-E** 

**NIDCR Grant Number:** 1U01DE027637

**UPenn IRB Number: 832750** 

Principal Investigator: Patricia Corby, DDS, MS

Sub-Investigator: Alexander Lin, MD

NIDCR Program Official: Dena Fischer, DDS, MSD, MS NIDCR Medical Monitor: Kevin McBryde, MD

4 January 2022

Version 11

## STATEMENT OF COMPLIANCE

The study will be conducted in accordance with the International Council for Harmonisation guidelines for Good Clinical Practice (ICH E6), the Code of Federal Regulations on the Protection of Human Subjects (45 CFR Part 46), and the NIDCR Clinical Terms of Award. All personnel involved in the conduct of this study have completed human subjects protection training.

### SIGNATURE PAGE

The signature below constitutes the approval of this protocol and the attachments provides the necessary assurances that this trial will be conducted according to all stipulations of the protocol, including all statements regarding confidentiality, and according to local legal and regulatory requirements and applicable US federal regulations and ICH guidelines.

Principal Investigator or Clinical Site Investigator:

Signed: Date: January 19, 2022

Name: Dr. Patricia Corby

Title: Principal Investigator

Signed:

Rlar dia Date: January 19, 2022

Name: Dr. Alexander Lin

Title: Co-Principal Investigator

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| | | GNATURE PAGE | |
| | | ABLE OF CONTENTSST OF ABBREVIATIONS | |
| | | ROTOCOL SUMMARY | |
| 1. | KEY | ROLES AND CONTACT INFORMATION | 12 |
| 2. | BAC | CKGROUND AND SCIENTIFIC RATIONALE | 13 |
| | 2.1. | BACKGROUND INFORMATION | |
| | 2.2. | PRELIMINARY DATA | 13 |
| | 2.3. | RATIONALE | |
| | 2.4. | STUDY POTENTIAL RISKS AND BENEFITS | 16 |
| | 2.4.1. | POTENTIAL RISKS | 16 |
| | 2.4.2. | POTENTIAL BENEFITS | 16 |
| 3. | OBJ | IECTIVES | 17 |
| | 3.1. | PRIMARY OBJECTIVE | |
| | 3.2. | SECONDARY OBJECTIVES | 17 |
| | 3.3. | EXPLORATORY OBJECTIVE | 17 |
| | 3.4. | STUDY OUTCOME MEASURES | 17 |
| | 3.4.1. | PRIMARY OUTCOME | 17 |
| | 3.4.2. | SECONDARY OUTCOMES | 18 |
| 4. | STU | DY DESIGN | 20 |
| 5. | STU | DY ENROLLMENT AND WITHDRAWAL | 21 |
| | 5.1. | SUBJECT INCLUSION CRITERIA | |
| | 5.2. | SUBJECT EXCLUSION CRITERIA | 21 |
| | 5.3. | STRATEGIES FOR RECRUITMENT AND RETENTION | |
| | DSMB | RECOMMENDATIONS REGARDING ENROLLMENT (12/10/2020): | 25 |
| | 5.4. | TREATMENT ASSIGNMENT AND RANDOMIZATION PROCEDURES | |
| | 5.5. | BLINDING PROCEDURES | |
| | 5.6. | SUBJECT WITHDRAWAL | 26 |
| | 5.6.1. | HANDLING OF SUBJECT WITHDRAWALS OR SUBJECT DISCONTINUATION OF STUDY | |
| | | ENTION | |
| | 5.7. | PREMATURE TERMINATION OR SUSPENSION OF STUDY | |
| 6. | | DY INTERVENTION | |
| | | STUDY PROCEDURAL INTERVENTION DESCRIPTION | |
| | 6.2. | ADMINISTRATION OF PROCEDURAL INTERVENTION | 28 |
| | 6.3. | PROCEDURES FOR TRAINING OF CLINICIANS ON PROCEDURAL INTERVENTION AND | |
| | | ORING TREATMENT FIDELITY | |
| | 6.4. | ASSESSMENT OF SUBJECT COMPLIANCE WITH STUDY PROCEDURAL INTERVENTION | |
| | 6.5. | CONCOMITANT MEDICATIONS/TREATMENTS AND REFERRALS FOR CARE | 29 |
| 7. | STU | DY SCHEDULE | 31 |
| | 7.1. | SCREENING AND BASELINE (SCREENING: DAY -60 TO -1; BASELINE: DAY -21 TO -1 | |
| | | VE TO INTERVENTION VISIT 1) | |
| | 7.2. | INTERVENTION VISITS (VISITS 1, 3, 5, 7, 9) | |
| | 7.3. | INTERVENTION VISITS (VISITS 2, 4, 6, 8) | 33 |
| | 7.4. | POST-INTERVENTION VISIT – FOLLOW UP VISIT (DAY 86+/- 7 DAYS) | 34 |
| | 7.5. | POST-INTERVENTION VISIT – FINAL STUDY VISIT (DAY 140 +/- 21 DAYS) | |
| | 7.6. | CLINICAL FOLLOW-UP | 35 |

| | 7.7.<br>7.8. | WITHDRAWAL VISIT | |
|---|---|---|---|
| | 7.9. | MISSED VISIT | 35 |
| 8. | OVE | RVIEW OF STUDY PROCEDURES/EVALUATIONS | 37 |
| | 8.1. | STUDY PROCEDURES/EVALUATIONS | |
| | 8.2. | QUESTIONNAIRES | 38 |
| | 8.3. | BLOOD DRAW | |
| | 8.4. | LABORATORY PROCEDURES/EVALUATIONS | |
| | | SPECIAL ASSAYS OR PROCEDURES | |
| | | SPECIMEN PREPARATION, HANDLING, AND STORAGE | |
| | 8.4.3. | | |
| | 8.5. | BIOBANKING FOR FUTURE RESEARCH | |
| | | STORAGE AND CONFIDENTIALITY OF SAMPLES | |
| | 8.5.2. | WITHDRAWAL OF SAMPLES | 40 |
| 9. | ASS | SESSMENT OF SAFETY | 41 |
| | 9.1. | SPECIFICATION OF SAFETY PARAMETERS | 41 |
| | 9.1.1. | UNANTICIPATED PROBLEMS | 41 |
| | 9.1.2. | ADVERSE EVENTS | 41 |
| | 9.1.3. | SERIOUS ADVERSE EVENTS | |
| | 9.2. | TIME PERIOD AND FREQUENCY FOR EVENT ASSESSMENT AND FOLLOW-UP | |
| | 9.3. | CHARACTERISTICS OF AN ADVERSE EVENT | |
| | 9.3.1. | | |
| | 9.3.2. | | |
| | 9.3.3. | | |
| | 9.4. | UNANTICIPATED PROBLEM REPORTING | |
| | 9.5. | SERIOUS ADVERSE EVENT REPORTING | |
| | 9.6. | HALTING RULES | 44 |
| 10 | ). STU | DY OVERSIGHT | 45 |
| 11 | I. CLII | NICAL SITE MONITORING | 46 |
| 12 | STA | TISTICAL CONSIDERATIONS | 47 |
| • | | STUDY HYPOTHESES | |
| | | SAMPLE SIZE CONSIDERATIONS | |
| | | PLANNED INTERIM ANALYSES | |
| | | SAFETY REVIEW | |
| | 12.4. | Analysis Plan | 49 |
| 13 | B. SOL | JRCE DOCUMENTS AND ACCESS TO SOURCE DATA/DOCUMENTS | 51 |
| | | ALITY CONTROL AND QUALITY ASSURANCE | |
| ' | | STAFF TRAINING | |
| | | VISIT-LEVEL QUALITY CONTROL | |
| | | CASE REPORT FORMS | |
| | | BIOSPECIMENS | |
| | | SEMIANNUAL QUALITY CONTROL | |
| 1 | | IICS/PROTECTION OF HUMAN SUBJECTS | |
| | | ETHICAL STANDARD | |
| | | INSTITUTIONAL REVIEW BOARD | |
| | | INFORMED CONSENT PROCESS | |
| | 15.4. | EXCLUSION OF WOMEN, MINORITIES, AND CHILDREN (SPECIAL POPULATIONS) | 55 |

| 15.6. | SUBJECT CONFIDENTIALITY CERTIFICATE OF CONFIDENTIALITY FUTURE USE OF STORED SPECIMENS AND OTHER IDENTIFIABLE DATA | 57 |
|---|---|---|
| 16. DA | TA HANDLING AND RECORD KEEPING | 58 |
| 16.1. | DATA MANAGEMENT RESPONSIBILITIES | 58 |
| 16.2. | DATA CAPTURE METHODS | 58 |
| | TYPES OF DATA | |
| 16.4. | SCHEDULE AND CONTENT OF REPORTS | 58 |
| 16.5. | STUDY RECORDS RETENTION | 59 |
| 16.6. | PROTOCOL DEVIATIONS | 59 |
| 16.7. | PUBLICATION/DATA SHARING POLICY | 59 |
| 17. LIT | ERATURE REFERENCES | 61 |
| | PPENDICES | |

#### LIST OF ABBREVIATIONS

ADL Activities of Daily Living

AE Adverse Event/Adverse Experience

American Joint Committee on Cancer - TNM Classification of Malignant

AJCC - TNM Tumors

ANC Absolute Neutrophil Count

ARMOR Commensal Oral Microbiota as a Trigger of Oral Mucositis Severity

CBC Complete Blood Count testing

CFR Code of Federal Regulations

chemoRT Chemoradiation therapy
CMP Clinical Monitoring Plan

CROMS Clinical Research Operations and Management Support

CTCAE Common Terminology Criteria for Adverse Events

CQMP Clinical Quality Management Plan

DHHS Department of Health and Human Services

DSMB Data and Safety Monitoring Board

EORTC QLQ- European Organization for Research and Treatment of Cancer Quality of

C-30 Life Questionnaire

EORTC QLQ- European Organization for Research and Treatment of Cancer Quality of

H&N35 Life Questionnaire with the additional Head & Neck specific module

FDA Food and Drug Administration

GCP Good Clinical Practice

GEE General Estimating Equation

H&N Head and Neck

HIV Human Immunodeficiency Virus

HNSCCs Head and Neck Squamous Cell Carcinomas

ICH International Council for Harmonisation

IMRT Intensity-modulated radiation therapy

IRB Institutional Review Board

Multinational Association of Supportive Care in Cancer and International

MASCC/ISOO Society of Oral Oncology

MOP Manual of Procedures

MSD MesoScale Discovery

NIDCR National Institute of Dental and Craniofacial Research, NIH, DHHS

NIH National Institutes of Health

NYU New York University

UPenn University of Pennsylvania, School of Dental Medicine

OCTOM Office of Clinical Trials Operations and Management

OHRP Office for Human Research Protections

OM Oral Mucositis

OMDP-IG Oral Mucosal Deterging and Dental Prophylaxis (Intervention Group)

PHI Protected Health Information

PI Principal Investigator

QM Quality Management

QOL Quality of life

RT Radiation Therapy

SAE Serious Adverse Event/Serious Adverse Experience

SOC-OH Standard of Care Oral Hygiene (Control Group)

SOC Standard of Care

US United States

WHO World Health Organization

#### PROTOCOL SUMMARY

**Title:** The ARMOR Trial: Commensal Oral Microbiota as a Trigger of Oral Mucositis Severity

**Précis:** This is a prospective, single blind, two arm, randomized, controlled trial to test the efficacy of an oral care protocol to treat oral mucositis (OM) in patients receiving radiation (RT) or chemoradiation (chemoRT) for head and neck cancer. This trial will also measure salivary proinflammatory cytokines, and evaluate other clinical effects of the intervention during cancer therapy. In addition, oral mucosal swabs will be collected for the future characterization of changes in the microbiome associated with OM severity.

Patients will be randomized in a 1:1 ratio to two different oral care protocols within 4 strata defined by type of RT (Proton beam therapy (Protons)) vs intensity-modulated radiation therapy (IMRT) and cancer treatment (RT versus chemoRT). Eligible subjects will be assigned to receive either the **Oral Mucosal Deterging and Dental Prophylaxis** protocol (OMDP) or a **Standard of Care Oral Hygiene** protocol (SOC-OH). Prior to randomization, all enrolled subjects will receive a baseline dental prophylaxis and fluoride varnish application prior to start of RT or chemoRT to ensure that all subjects enter the study with comparable oral health. **Subjects assigned to OMDP** will receive the OMDP Protocol (*Oral Mucosal Deterging and Dental Prophylaxis*) at weekly intervention visits. **Subjects randomized to the SOC-OH** will receive oral health instructions following the *American Dental Association Guidelines*<sup>1</sup> and will have their teeth cleaned (brushed) during weekly intervention visits; no treatment to the oral mucosa will be provided to this group.

At each bi-weekly study visit, study assessments will include the collection of saliva and oral mucosal swabs, an oral exam and OM assessment, and the completion of questionnaires. During the course of the study, subjects will attend one baseline visit, up to 9 intervention visits, and follow-up visits approximately 1 month and 3 months after completion of RT. Local supportive care, including normal saline rinses, topical anesthetics, mixed medication mouthwashes (e.g. Magic Mouthwash), feeding tubes, and pain management will be allowed according to each recruitment site's standard of care procedures.

# **Objectives:**

<u>Primary Objective:</u> To test the efficacy of the OMDP protocol compared to SOC-OH on OM severity in head and neck cancer patients undergoing RT or chemoRT.

The primary outcome measure is OM severity as measured by the World Health Organization's Oral Toxicity Scale (WHO OTS).

# **Secondary Objectives:**

- 1) To compare changes in salivary **proinflammatory cytokines** between the OMDP and SOC-OH groups.
- 2) To evaluate differences between the OMDP and SOC-OH groups in the following clinical indicators: a) duration of and time to onset of severe OM, b) salivary hypofunction, c) average mouth and throat soreness [MTS], and d) quality of life and function [EORTC QLQ 30 and EORTC QLQ HN35].

The secondary outcome measures are changes in: salivary proinflammatory cytokines, duration and time to onset of severe OM, OM severity as measured by the Common Terminology Criteria for Adverse Events (CTCAE), salivary hypofunction, symptoms, quality of life, and function.

Exploratory Objective. To estimate progression-free survival and overall survival by intervention group.

The central hypothesis is that a weekly regimen of targeted professional oral care during anti-cancer treatment prevents harmful ecological shifts in the oral cavity and consequently reduces the duration and severity of OM, reduces OM local inflammation, and improves oral health, thereby improving overall quality of life during cancer treatment. The rationale is that the cleansing of dead, damaged, or infected oral mucosa tissues in combination with mechanical removal of dental plaque and calculus in the oral cavity to facilitate biofilm disruption and endotoxin flushing during RT/chemoRT treatment, improves the healing potential of the oral tissues and suppresses OM severity.

## Population:

A total of 120 male and female subjects (N=120) aged 18 years and older who will undergo different modalities of RT [IMRT or Protons] with or without combined chemotherapy for head and neck cancer will be enrolled.

Phase:

Ш

Clinical Hospital of the University of Pennsylvania Center (s): Perelman Center for Advanced Medicine

3400 Civic Center Blvd Philadelphia, PA 19104

Perelman School of Medicine, University of Pennsylvania

Department of Oral & Maxillofacial Surgery Perelman Center for Advanced Medicine

3400 Civic Center Blvd., 4th Floor South Pavilion

Philadelphia, PA 19104

School of Dental Medicine, University of Pennsylvania

Number of Two core laboratories: Core The Forsyth Institute

Laboratories: National Institute of Nursing Research (NINR)

Statistical Center:

NYU Langone Health, School of Medicine

Description of Intervention:

The study intervention will consist of weekly visits during which a dental professional will administer the OMDP intervention protocol. The OMDP comprises a professional dental prophylaxis including periodontal surface debridement (a light-touch, gentle form of instrumentation performed with an ultrasonic instrument to promote plaque removal, to facilitate biofilm disruption and endotoxin flushing, but yet with the preservation of the periodontal cementum) followed by cleansing and deterging of the oral mucosal surfaces using a soft bristled manual toothbrush and a deterging agent.

The standard of care intervention for the control group will consist of weekly visits at which subjects will receive oral health instructions and have their teeth brushed.

Study Duration:

Approximately 5 years

Subject
Participation
Duration:

Approximately 5 months

Estimated Appro

Approximately 3.5 years

Complete Enrollment:

### SCHEMATIC OF STUDY DESIGN:

Screening (Day -60 to -1) Baseline (Day -21 to -1) Must occur prior to randomization.

A. Obtain informed consent. Screen potential subjects by inclusion and exclusion criteria, obtain history, vital signs, oral exam.

\*B. Saliva and oral swab collection, questionnaires, perio assessment, dental prophylaxis. Blood draw\*\*.

Screening and Baseline can happen at the same visit, however

\*Assessments in "B" must be done within the Baseline window.

\*\*Blood draw may occur any time prior to the start of RT.

VISIT 1 (Day 0, up to 5 days after the start of RT

Randomization - AEs, oral exam, mucositis assessment, saliva, and oral swab collection, questionnaires, study intervention.



VISIT 3 (Day  $14 \pm 3$  days)

questionnaires, study intervention.

VISIT 4 (Day 21 ± 3 days)

Study intervention and mucositis assessment

VISIT 5 (Day 28 ± 3 days)

AEs, oral exam, mucositis assessment, saliva and oral swab collection, questionnaires, study intervention.

VISIT 6 (Day 35 ± 3 days)

Study intervention and mucositis assessment

**VISIT 7 (Day 42 (± 3 days)** 

AEs, oral exam, mucositis assessment, saliva and oral swab collection, questionnaires, study intervention.

VISIT 8 (Day 49  $\pm$  3 days)

Study intervention and mucositis assessment

VISIT 9 (Day  $56 \pm 3$  days)

AEs, oral exam, mucositis assessment, saliva and oral swab collection, questionnaires, study intervention.

VISIT 10 (Day 86 ± 7 days)

AEs, oral exam, mucositis assessment

**POST RT VISIT** 

Visit 11 (Day 140 ± 21 days)

AEs, oral exam (including perio assessment), saliva and oral swab collection, questionnaires, study intervention if needed.

## 1. KEY ROLES AND CONTACT INFORMATION

**Program Principal** 

Patricia Corby, DDS, MS Investigator Associate Dean for Translational Research

**Contact PI** Associate Professor

Department of Oral Medicine

University of Pennsylvania School of Dental Medicine

Email: patcorby@UPenn.edu

Phone: 215-898-1162 240 South 40th Street Philadelphia, PA 19104

**Program Co-Principal** Investigator

Alexander Lin, M.D. Associate Professor

Vice Chair of Faculty Affairs

Chief, Head and Neck Cancer Section

Medical Director, Roberts Proton Therapy Center

Department of Radiation Oncology

Perelman School of Medicine, University of Pennsylvania

Email: alexander.lin@uphs.UPenn.edu

Fax: 215-349-5445 Phone: 215-662-3198

**NIDCR Medical** 

**Monitor:** 

Kevin McBryde, MD NIH/NIDCR/DER

6701 Democracy Boulevard, Room 638

Bethesda, MD 20892-4878 Phone: 301 594 0170

Email: mcbrydekd@mail.nih.gov

**NIDCR Program** 

Dena Fischer, DDS, MDS, MS

Official: National Institute of Dental and Craniofacial Research/NIH

6701 Democracy Blvd, MSC 4878

Bethesda, MD 20892-4878 Phone: (301) 594-4876 Email: dena.fischer@nih.gov